CLINICAL TRIAL: NCT05486611
Title: A Randomized Controlled Trial of a Digital Therapeutic (WB002) and Educational App (ED002) for Depression Among Adolescents
Brief Title: Digital Therapeutic vs Educational App for Depression Among Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to difficulty enrolling patients in the proposed time frame
Sponsor: Woebot Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W-GenZD-004
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Depression
Keywords: Mental Health; Adolescent; Digital Therapeutic; Chatbot; Mental Health App
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-GenZD Mobile Application Group (Experimental): Participants assigned to the W-GenZD mobile application group will be asked to download and use the W-GenZD mobile application that will provide information and tools through a chatbot (a computer program designed to communicate with users). Participants will be invited to use the mobile application as often as they like during the 4-week treatment period - we will encourage 5 to 10 minutes of daily use.
  Interventions: Device: W-GenZD Mobile Application
- Digital Education Application Group (Sham Comparator): Participants assigned to the Digital Education mobile app group will be given instructions on how to download and access the application that will provide general health information. A new article will be provided to the participant at a rate of once per week across the 4 weeks (4 articles total) and they will receive a weekly notification when a new article is available. Each article will be available for one week from release date. We expect a target dosage of roughly 30 minutes per week (120 min), which would make it comparable to Woebot (about 5 min per day X 28 days = 140 min).
  Interventions: Device: Digital Education Application (W-EdZD)

INTERVENTIONS:
Device: W-GenZD Mobile Application — W-GenZD is a mobile application program that delivers evidence-based therapy for the symptoms of mild-moderate depression and anxiety in adolescents in brief "conversations" with a fully automated relational agent called Woebot. It is a brief, self-guided 4 week-intervention that draws from cognitive behavioral therapy (CBT), interpersonal psychotherapy for adolescents (IPT-A), and elements of dialectical behavior therapy (DBT), depending on the presenting situation, to help the adolescent develop emotion regulation skills in the context of their everyday life. In this way, the mobile application is designed to be targeted, relevant, and integrated into the lived experience of adolescents, capable of delivering the appropriate technique for the problem at hand, at the time of need.
  Arms: W-GenZD Mobile Application Group
Device: Digital Education Application (W-EdZD) — Digital Education will be available to the participant via the 'Quest GenZ' smartphone application but will be devoid of active elements included in WB002. We will source this material from kidshealth.org, which is supported by Nemours Children's Health. We have received permission to use their content.
  The materials are written at an 8th grade reading level and will include general health (e.g., food plate guide, caffeine, online safety, study skills) articles. A new article will be provided to the participant at a rate of once per week across the 4 weeks (4 articles total) and they will receive a weekly notification when a new article is available. Each article will be available for one week from release date.
  Arms: Digital Education Application Group

SUMMARY:
The primary aim of this study is to investigate the difference in depression symptoms at 4-weeks across two types of programs for addressing depressive symptoms, including Woebot (WB002) and Digital Education (ED002). The secondary aim of this study is to investigate the difference in anxiety symptoms at 4-weeks across the two programs. The tertiary aim of this study is to evaluate the feasibility, acceptability, and satisfaction of each program.

ELIGIBILITY:
Inclusion Criteria:

1. Be 13-17.5 years of age
2. Be a U.S. Resident
3. Able to read and write in English
4. If currently on medication: regular, stable dose of antidepressant medications (e.g., escitalopram/Lexapro, fluoxetine/Prozac) for at least 60 days at screening
5. If currently receiving psychotherapy: must be in therapy for at least 4 weeks at screening
6. Own or have regular access to a smartphone (operating systems: Android 6 or later and iOS 13 or later) that can receive SMS messages, and has reliable Wi-Fi access or sufficient data to engage with study app
7. Available and committed to engage with the program for a 8-week duration and complete assessments
8. Participants must be able to understand and willing to provide informed assent and to comply with all study procedures and restrictions
9. Willingness to provide parent/guardian contact information to provide eConsent and participate in clinical interviews

Exclusion Criteria:

1. PHQ-A score less than 10
2. Lifetime diagnosis of a psychotic disorder (including schizophrenia or schizoaffective disorder)
3. Lifetime diagnosis of bipolar disorder
4. Lifetime diagnosis of autism spectrum disorder or pervasive developmental disorder (e.g., Asperger syndrome, Rett's syndrome, or pervasive developmental disorder not otherwise specified)
5. Current (past year) diagnosis of a substance use disorder
6. Suicide attempt or suicidal ideation with plan and intent within the past 12 months
7. Previous Woebot application use
8. Enrollment of more than one member of the same household

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire for Teens (PHQ-A) | Change from Screening to Mid-treatment at 2 weeks; Change from Screening to Post-treatment at 4 weeks; Change from Screening to Follow-up at 6 and 8 weeks
  Measure of depression severity. An 8-item abbreviated version of the PHQ-9 used to assess mood and anxiety symptoms respectively. The PHQ-8 excludes an item assessing suicidality. Total score between 0-27, where higher scores indicate greater levels of depression.

SECONDARY OUTCOMES:
General Anxiety Disorder Questionnaire (GAD-7) | Change from Baseline to Mid-treatment at 2 weeks; Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to Follow-up at 6 and 8 weeks
  Measure of anxiety. A 7-item brief self-report measure used to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. Total score between 0-21, where higher scores indicate greater levels of anxiety.
Children's Depression Rating Scale-Revised (CDRS-R) | Change from Baseline to Post-treatment at 4 weeks
  Measure of depression. The CDRS-R is a brief rating scale based on a semi-structured interview with the child. Designed for 6- to 12-year-olds, it has been successfully used with adolescents. Seventeen symptom areas are assessed during the interview with a 5- to 7-point rating scale: Impaired Schoolwork, Difficulty Having Fun, Social Withdrawal, Appetite Disturbance, Sleep Disturbance, Excessive Fatigue, Physical Complaints, Irritability, Excessive Guilt, Low Self-Esteem, Depressed Feelings, Morbid Ideation, Suicidal Ideation, Excessive Weeping, Depressed Facial Affect, Listless Speech, and Hypoactivity. Total scores range from 17- 113. A score of ≥40 is indicative of depression, whereas a score ≤28 is often used to define remission (minimal or no symptoms).
PROMIS Pediatric Global Health (PGH-7) | Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to Follow-up at 8 weeks
  Measure of global health. A 7-item self-report measure of a child's global health developed for children and adolescents in the 8-17 age range. Items assess general, physical, mental, and social health, with response options on a 5-point likert scale. Total score ranges from 1-35, where higher scores indicate better health.
Client Satisfaction Questionnaire (CSQ-8) | Post-treatment at 4 weeks
  An 8-item measure used to assess client's satisfaction with treatment on a 4-point scale (1 = "very dissatisfied" to 4 = "very satisfied"). Example questions include, "How would you rate the quality of service you received"? and "Did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with the W-GenZD mobile application or the W-EdZD mobile application.
Usage Rating Profile - Intervention (URPI)-Feasibility | Post-treatment at 4 weeks
  Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Responses range from 1 = "slightly disagree" to 6 = "strongly agree". Scores are averages, with greater scores indicating greater intervention feasibility.
Usage Rating Profile - Intervention (URPI)-Acceptability | Post-treatment at 4 weeks
  Measure of acceptability. A 6-item subscale that inquires about intervention acceptability. Responses range from 1 = "slightly disagree" to 6 = "strongly agree". Scores are averages, with greater scores indicating greater intervention acceptability.
Working Alliance Inventory - Short Revised (WAI-SR) | Day 4; Change from Day 4 to Post-treatment at 4 weeks
  Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Scores range from 5-20, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot" for participants randomized to the W-GenZD treatment arm.
Alexithymia Questionnaire for Children (AQC) | Change from Baseline to Day 4; Change from Baseline to Post-treatment at 4 weeks
  Measure of the alexithymia construct. A self-report questionnaire based on the original Toronto Alexithymia Scale (TAS-20), revised with language oriented toward children and adolescents. A total of 20 items comprises the AQC, with responses on a 3-point Likert-scale (ranging from 0 = not true to 2 = often true). The AQC measures 3 core factors including difficulty identifying feelings (7 items), difficulty describing feelings (5 items), and externally-oriented thinking (8 items). Higher total scores correspond to an elevated presence of the factor. Emotional awareness can be measured using the 12 items that make up the difficulty identifying feelings and difficulty describing feelings factors, so we will be administering these subscales.
Cognitive Flexibility Inventory (CFI) | Change from Baseline to Post-treatment at 4 weeks
  Measure of cognitive flexibility. A 20-item assessment designed to measure three aspects of cognitive flexibility: the tendency to perceive difficult situations as controllable; the ability to perceive multiple alternative explanations for life occurrences and human behavior; and the ability to generate multiple alternative solutions to difficult situations. Total scores range from 7-140, with Alternatives scale ranging from 7-91 and Control scale from 7-49. There are currently no established cutoff scores for high, moderate, and low flexibility across the scales, though higher scores indicate greater flexibility.
CAR, RELAX, ALONE, FORGET, FRIENDS, TROUBLE (CRAFFT) | Baseline
  Measure of substance use. A validated 9-item screening tool designed to identify substance use past 12 months, substance-related risk, and substance use disorder in adolescents aged 12-21. Total CRAFFT scores range from 0-6, where a score of 0 indicates low risk level, a score <2 is medium risk, and a score >= 2 is deemed high risk.
Woebot Reflection Questionnaire (WRQ) | Change from Baseline to Post-treatment at 4 weeks; Change from Baseline to Follow-up at 8 weeks
  Measure of user perceptions on three domains: symptoms, abilities, and quality of life. The 17-item measure assesses user perceptions on symptoms, abilities, and quality of life over the past 2 weeks. The Symptoms domain consists of 4-items asking the user to rate the severity of symptoms related to their mood, such as sadness, stress, irritability, and negative thoughts. The 7-item Abilities domain assesses how well users were able to copy, complete, or navigate responsibilities, activities, or emotions. The Quality of Life domain is 6-items and assesses the frequency of users experienced physical and social wellbeing. All responses are presented with Likert responses. This measure has not undergone psychometric testing and will be used in this study to evaluate its preliminary validity and sensitivity to change against more validated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Robinson, PhD, Principal Investigator — Woebot Health
Locations (1):
- Woebot Health, San Francisco, California, United States